CLINICAL TRIAL: NCT05011617
Title: Monitored Anesthesia Care Versus Intubated General Anesthesia for Open Heart Surgery Under Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ShuGuang Hospital (Other)
Responsible Party: Principal Investigator, Jiangang Song, Director of anesthesiology department of Shuguang Hospital, ShuGuang Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 81603450
Record Dates: First submitted 2021-08-08; First posted 2021-08-18 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Monitored Anesthesia Care; Cardiac Surgery; Postoperative Recovery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: We set a blind code in case patients have adverse effects. The random code and blind code will be conducted using opaque envelopes by a "third party" independent of the study. The envelopes will be sealed and shuffled, and the assignment records will not be disclosed until the end of the study. Trial participants, cardiothoracic surgeons, anesthesiologists, outcome assessors, and data analysts will be blinded to the treatment allocation to minimize potential sources of bias. Only the nurse of the anesthesiology department (having received specialized acupuncture training) will know the participants' group allocations. However, this nurse will not know any other information about the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAC group (Experimental): Electroacupuncture was performed for two consecutive days before surgery (2 daily 30-min sessions) by a licensed acupuncturist at 4.0 mA using an alternating frequency of 2 and 100 Hz (every 1.5 seconds) (LH-202, Huawei, Beijing, China). Acupoints included bilateral Yunmen (LU2), Zhongfu (LU1), Lieque (LU7), and Neiguan (PC6). On the day of surgery, electroacupuncture started upon the completion of a loading dose of dexmedetomidine, was suspended when CPB started (to avoid interference with electrocardiogram recording) and continued until the end of surgery.
  Interventions: Device: Non-intubation and monitoring anesthesia care (MAC)
- IGA group (No Intervention): Anesthesia was induced with propofol (2.0-3.5 μg/mL) by target control infusion and 0.3-0.5 μg/kg sufentanil. Tracheal intubation was facilitated by rocuronium (1.0 mg/kg). Anesthesia was maintained using isoflurane at 0.7-1.0 minimal alveolar concentration in a gas mixture of oxygen and air and remifentanil (0.05-0.2 μg·kg-1·min-1) by intravenous injection pump. Sufentanil dose was totally 2.5-4.0 μg/kg. Muscle relaxation was achieved using 1/3-1/4 of the induction dose every 40-60 min based on a train of four. Mechanical ventilation with 80% O2 in air was used. Tidal volume (7-8 mL/kg) and respiratory rate (10-12/min) were adjusted according to PETCO2 to achieve normal ventilation (PETCO2 35-45 mmHg).

INTERVENTIONS:
Device: Non-intubation and monitoring anesthesia care (MAC) — Non-intubation and monitoring anesthesia care (MAC) consisted of non-intubation technique, local anesthesia at the site of sternotomy, sedation with dexmedetomidine, analgesia with remifentanil/sufentanil, and electroacupuncture.
  Arms: MAC group

SUMMARY:
Though Cardiac surgery under cardiopulmonary bypass (CPB) under epidural anesthesia in conscious patients is associated with increased risk of epidural hematoma. The investigators developed a monitored anesthesia care (MAC) platform for cardiac surgery under CPB. In the current prospective study, the investigators investigated the safety and effectiveness of the MAC platform versus intubated general anesthesia (IGA) in patients receiving elective open-heart surgery.

The study included adult patients who were scheduled to undergo open-heart surgery under CPB at Shuguang Hospital between April 2012 and December 2021. MAC consisted of local anesthesia at the site of sternotomy, sedation with dexmedetomidine, analgesia with remifentanil/sufentanil and electroacupuncture. MAC versus IGA was chosen by the patients. The investigators will investigate the safety and effectiveness of the MAC platform versus IGA in patients receiving elective open-heart surgery.

DETAILED DESCRIPTION:
The detailed description of clinical trial will be published by protocol later.

ELIGIBILITY:
Inclusion Criteria:

* 1) NYHA class II or less;
* 2) expected aortic block time at ≤ 120 min;
* 3) body mass index (BMI) between 18 and 30 kg/cm2.

Exclusion Criteria:

* 1) systolic pulmonary blood pressure > 70 mmHg;
* 2) chronic obstructive pulmonary disease, obstructive sleep apnea syndrome, or simplified airway risk index > 3;
* 3) Child-Pugh grade B or C liver insufficiency or renal insufficiency (24-h creatinine clearance < 80 mL/min and blood urea nitrogen > 7.5 mmol/L);
* 4) coagulopathy (aPTT prolongation > 10 seconds versus normal controls, PT prolongation > 3 seconds versus normal controls, and INR > 3.0).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
intraoperative consumption of opioids | end of the surgery, up to 48 hours after surgery
  intraoperative consumption of sufentanil and remifentanil

SECONDARY OUTCOMES:
time to drinking | through study completion, an average of 24 hours
  The interval between the end of surgery and the first drink

OTHER OUTCOMES:
length of ICU stay | through study completion, an average of 12 days
  the length of time about transfer out of ICU after surgery
The Vasoactive-inotropic Score | end of the surgery, up to 48 hours after surgery
  The vasoactive-inotropic score was used to evaluate the dose of various vasoactive drugs and calculated by the following formula: Vasoactive-inotropic score = dopamine (×1) + dobutamine (×1) + amrinone (×1) + milrinone (×15) + epinephrine (×100) + norepinephrine (×100) + isoprenaline (×100). The minimum value was 0 and the maximum values had no upper limit. The higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jianggang Song, MD, Study Chair — Acupuncture and Anesthesia Research Institute, Shanghai, China
Locations (1):
- Shuguang Hospital of Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make IPD available. The results belong to the research team.